CLINICAL TRIAL: NCT00575783
Title: Impact of Hypoglycemia Unawareness on Brain Metabolism Cognition in T1DM
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Miami (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0505000077_B; R01DK072409 (NIH); HIC# 0505000077
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: type 1 diabetes; hypoglycemia; magnetic resonance imaging
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1A, 1B: Type 1 diabetic subjects with a history of severe hypoglycemia and hypoglycemia unawareness who:
  1A) meet criteria for islet cell transplantation and are referred by a participating islet cell transplantation center
  1B) meet similar criteria but are not currently planning islet cell transplantation
- 2: Type 1 diabetics who are not optimally controlled (>8% HbA1c) and rarely experience hypoglycemia
- 3: Healthy non-diabetics

SUMMARY:
The research study is designed to examine the impact of low blood sugar on brain function in individuals with Type 1 Diabetes who have frequent and severe hypoglycemia (low blood sugar) compared to those who do not.

DETAILED DESCRIPTION:
During the course of treating diabetes (for example, after an insulin injection), blood sugar levels will sometimes drop too low. This condition is known as hypoglycemia. Normally, a healthy body responds to hypoglycemia by producing a number of "anti-insulin" hormones which raise blood sugar levels. In addition, these hormones provide the individual with warning signals of hypoglycemia, including hunger, sweating, shaking and heart palpitations. These warning signals allow diabetics to correct low blood sugar levels by eating sugar tablets or by having a snack.

Unfortunately, and for unclear reasons, many people with longstanding diabetes lose their ability to recognize low blood sugar levels-a condition called "hypoglycemia unawareness." The brain, in particular, is extremely sensitive to hypoglycemia. Unable to sense and respond to low blood sugar levels, these individuals may experience a sudden onset of blurred vision, confusion, seizures, coma, or even death.

In recent years, a new technique called "islet cell transplantation" has been developed as an alternate means of treating insulin-dependent diabetes. Pancreatic islet cells (the cells that produce insulin), from human donors, are injected into the diabetic patient's liver where the cells are capable of making insulin and can regulate blood sugar levels without the need for insulin injections. Currently, this technique is used primarily in patients with severe hypoglycemia unawareness.

While it is known that islet cell transplantation can reduce the risk of severe hypoglycemia, the effects of transplantation on hypoglycemia unawareness are unknown. This study is designed to investigate why hypoglycemia unawareness happens and the impact it has on brain function in individuals with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for all subjects:

  * Age 18-49
  * > 85 kg
  * BMI <27female <28 male
  * able to provide written informed consent
  * able to speak and read English fluently
  * must meet Magnetic Resonance safety evaluation

Inclusion criteria for Group 1A:

* T1DM undergoing intensive clinical management and currently on the islet transplant list
* History of severe hypoglycemia

Inclusion criteria for Group 1B:

* T1DM undergoing intensive clinical management
* History of severe hypoglycemia unawareness

Inclusion criteria for Group 2:

* T1DM with poor glycemic control, HbA1c > 8%
* no episodes of hypoglycemia requiring assistance from another person for at least 1 yr, no episodes in last 4 weeks, and hypoglycemia aware

Exclusion Criteria:

Group 1A: (T1DM subjects being considered for islet cell transplantation)

* Detectable c-peptide level
* Untreated proliferative retinopathy
* Creatinine clearance < 65 ml/min/1.73 m2
* Serum creatinine ≥1.5 mg/dL
* Previous pancreas or islet transplant
* Positive pregnancy test, or presently breast-feeding, or failure to follow effective contraceptive measures
* Active infection including hepatitis C, hepatitis B, HIV, or TB (or under treatment for suspected TB ), or subjects with a positive PPD performed within 1 yr. of enrollment, and no history of adequate prophylaxis
* Invasive aspergillus infection within year prior to study entry
* Any history of malignancy except for adequately treated squamous or basal cell carcinoma of the skin
* Active alcohol or substance abuse- includes cigarette smoking (must be abstinent for 6 months)
* History of non-adherence to prescribed regimens
* Psychiatric disorder making the subject not a suitable candidate for transplantation
* Baseline Hgb < 10.5 g/dL in females, or < 13 g/dL in males; lymphopenia (<1,000/μL), or leukopenia (< 3,000 total leukocytes/μL), or an absolute CD4+ count < 500/μL
* History of coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after transplantation (low-dose aspirin treatment is allowed) or patient with INR >1.5
* Severe co-existing cardiac disease, as determined by referring center
* Baseline liver function tests outside of normal range (an initial liver function test panel with any values >1.5 times normal upper limits will exclude a patient without a re-test; a re-test for any values between normal and 1.5 times normal will be made, and if the values remain elevated above normal, the patient will be excluded), or history of significant liver disease
* Severe unremitting diarrhea or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications
* Addison's disease as determined by clinical history
* Under treatment for a medical condition requiring chronic use of systemic steroids
* Any medical condition or medication that, in the opinion of the investigators, will interfere with the safe completion of the study or study outcomes

Group 1 B: (T1DM with Severe Hypoglycemia Unawareness not on the Transplant List)

* Detectable C-peptide level
* Serum creatinine ≥1.5 mg/dL
* Positive pregnancy test, or presently breast-feeding, or failure to follow effective contraceptive measures
* Active alcohol or substance abuse- includes cigarette smoking (must be abstinent for 6 months)
* Psychiatric disorder making the subject not a suitable candidate for transplantation
* Baseline Hgb < 10.5 g/dL in females, or < 13 g/dL in males
* Baseline liver function tests outside of normal range (an initial liver function test panel with any values >1.5 times normal upper limits will exclude a patient without a re-test; a re-test for any values between normal and 1.5 times normal will be made, and if the values remain elevated above normal, the patient will be excluded), or history of significant liver disease
* Under treatment for a medical condition requiring chronic use of systemic steroids
* Any medical condition or medication that, in the opinion of the investigators, will interfere with the safe completion of the study or study outcomes

Group 2: (T1DM control subjects)

* Detectable C-peptide level
* Serum creatinine ≥1.5 mg/dL
* Positive pregnancy test, or presently breast-feeding, or failure to follow effective contraceptive measures
* Any history of malignancy except for adequately treated squamous or basal cell carcinoma of the skin
* Active alcohol or substance abuse- includes cigarette smoking (must be abstinent for 6 months)
* Baseline Hgb < 10.5 g/dL in females, or < 13 g/dL in males Baseline liver function tests outside of normal range (an initial liver function test panel with any values >1.5 times normal upper limits will exclude a patient without a re-test; a re-test for any values between normal and 1.5 times normal will be made, and if the values remain elevated above normal, the patient will be excluded), or history of significant liver disease
* Addison's disease as determined by clinical history
* Under treatment for a medical condition requiring chronic use of systemic steroids
* Any medical condition or medication that, in the opinion of the investigators, will interfere with the safe completion of the study or study outcomes

Group 3: (Normal Controls)

* FBG > 100 mg/dL
* Serum creatinine ≥1.5 mg/dL
* Positive pregnancy test, or presently breast-feeding, or failure to follow effective contraceptive measures
* Any history of malignancy except for adequately treated squamous or basal cell carcinoma of the skin
* Active alcohol or substance abuse- includes cigarette smoking (must be abstinent for 6 months)
* Baseline Hgb < 10.5 g/dL in females, or < 13 g/dL in males
* Baseline liver function tests outside of normal range (an initial liver function test panel with any values >1.5 times normal upper limits will exclude a patient without a re-test; a re-test for any values between normal and 1.5 times normal will be made, and if the values remain elevated above normal, the patient will be excluded), or history of significant liver disease
* Under treatment for a medical condition requiring chronic use of systemic steroids
* Any medical condition or medication that, in the opinion of the investigators, will interfere with the safe completion of the study or study outcomes

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group 1A) T1DM subjects with severe hypoglycemia unawareness and awaiting islet cell transplantation will be referred by participating islet transplantation centers.
  Group 1B) T1DM subjects with severe hypoglycemia unawareness but not awaiting islet cell transplantation will be from the greater New Haven, CT area.
  Group 2)T1DM, not optimally controlled and without hypoglycemia unawareness will be from the greater New Haven, CT area.
  Group 3) Non-Diabetics from the greater New Haven CT area.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2005-08; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- See also: American Diabetes Association — http://www.diabetes.org/
- See also: Juvenile Diabetes Research Foundation — http://www.jdrf.org/